CLINICAL TRIAL: NCT03795740
Title: The Precise Surgical Treatment of Chronic Thromboembolic Pulmonary Hypertension: Pulmonary Endarterectomy Guided by Three-dimensional Pulmonary Angiography
Brief Title: Pulmonary Endarterectomy Guided by CT Scanning for Patients With Chronic Thromboembolic Pulmonary Hypertension----PEACT
Acronym: PEACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheng Liu (Other)
Responsible Party: Sponsor-Investigator, Sheng Liu, Adult Cardiac Surgery Center, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: liusheng-1999
Record Dates: First submitted 2018-12-19; First posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension; Pulmonary Embolism
Keywords: computed tomography; chronic thromboembolic pulmonary hypertension; pulmonary endarterectomy; result; randomized controlled trial
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Precise (Experimental): precise PEA therapy with the guide of 3-D imaging techniques
  Interventions: Diagnostic Test: 3-D CT scanning
- Placebo (Placebo Comparator): traditional PEA therapy solely by surgical probe and traditional CT scanning/pulmonary angiography method
  Interventions: Diagnostic Test: 3-D CT scanning

INTERVENTIONS:
Diagnostic Test: 3-D CT scanning — For patients in Group 1,precisely analyzed CT scanning and/or pulmonary angiography will be done,and the patients in Group 1 will receive PEA procedure with the guide of precise 3-D imaging techniques

SUMMARY:
This study is a effectiveness study of the application of high-definition enhanced computed-tomography for patients with chronic thromboembolic pulmonary hypertension(CTEPH).The patients with CTEPH was randomized into 2 groups,precise pulmonary endarterectomy group(guided by enhanced CT scanning) and traditional pulmonary endarterectomy group,the hemodynamic changes tested with right sided heart catherization from baseline to post-operative period and end-point including peri-operative deaths,follow-up mortality,follow-up parameters of ultrasonic cardiogram(UCG),right-sided heart catherization(RHC),nuclear magnetic resonance imaging(MRI),cardiac pulmonary exercise test(CPET) are documented,so as to compare the prognosis between these 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosed with chronic thromboembolic pulmonary hypertension with the right-sided cathrization and pulmonary angiography;
* The computed tomography imaging implied that the location of the embolism could be reached with surgeries;

Exclusion Criteria:

* Beyond the age limit described above,or combined with other severe conditions such as severe organ dysfunction and considered contraindicated for surgical therapy by the cardiac surgeons;
* Without the consent by the patient or his/her families;
* Acute pulmonary embolism;
* Pulmonary sarcoma;
* Pulmonary arteritis;
* Combined with cardiogenic pulmonary hypertension or idiopathic pulmonary hypertension;

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline pulmonary systolic pressure within 1 month | within 1 month before and after pulmonary endarterectomy surgery
  Systolic pulmonary pressure result tested by right-sided heart
Change from Baseline pulmonary mean pressure within 1 month | within 1 month before and after pulmonary endarterectomy surgery
  Mean pulmonary pressure result tested by right-sided heart
Change from Baseline pulmonary vascular resistance within 1 month | within 1 month before and after pulmonary endarterectomy surgery
  Pulmonary vascular resistance result tested by right-sided heart
Change from Baseline cardiac output within 1 month | within 1 month before and after pulmonary endarterectomy surgery
  Cardiac output result tested by right-sided heart
mortality rate after surgery | immediately after the surgery to the longest 48 months follow-up period
  mortality rate after surgery

SECONDARY OUTCOMES:
Follow-up right ventricular ejection fraction | 3-24 months after the surgeries
  Assessed by UCG
Follow-up tricuspid annular plane systolic excursion | 3-24 months after the surgeries
  Assessed by UCG
Follow-up right ventricular anterior-posterior diameter | 3-24 months after the surgeries
  Assessed by UCG
Follow-up tricuspid insufficiency level | 3-24 months after the surgeries
  Assessed by UCG
Follow-up peak oxygen consumption (Peak O2) result | 6-24 months after the surgeries
  Assessed by cardio-pulmonary exercise test (CPET)
Follow-up Peak O2% | 6-24 months after the surgeries
  Assessed by CPET
Follow-up 6-minutes walking distance | 6-24 months after the surgeries
  Assessed by CPET
follow-up NYHA classes | 6-24 months after surgeries
  NYHA classes in the follow up period,either with telephone follow-up or out-patient follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital,Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
We have yet no plan to share IPD with other researchers

REFERENCES:
- [Background] Jamieson SW, Kapelanski DP, Sakakibara N, Manecke GR, Thistlethwaite PA, Kerr KM, Channick RN, Fedullo PF, Auger WR. Pulmonary endarterectomy: experience and lessons learned in 1,500 cases. Ann Thorac Surg. 2003 Nov;76(5):1457-62; discussion 1462-4. doi: 10.1016/s0003-4975(03)00828-2. PMID 14602267
- [Background] Pengo V, Lensing AW, Prins MH, Marchiori A, Davidson BL, Tiozzo F, Albanese P, Biasiolo A, Pegoraro C, Iliceto S, Prandoni P; Thromboembolic Pulmonary Hypertension Study Group. Incidence of chronic thromboembolic pulmonary hypertension after pulmonary embolism. N Engl J Med. 2004 May 27;350(22):2257-64. doi: 10.1056/NEJMoa032274. PMID 15163775
- [Background] Coquoz N, Weilenmann D, Stolz D, Popov V, Azzola A, Fellrath JM, Stricker H, Pagnamenta A, Ott S, Ulrich S, Gyorik S, Pasquier J, Aubert JD. Multicentre observational screening survey for the detection of CTEPH following pulmonary embolism. Eur Respir J. 2018 Apr 4;51(4):1702505. doi: 10.1183/13993003.02505-2017. Print 2018 Apr. PMID 29563171
- [Background] Kirson NY, Birnbaum HG, Ivanova JI, Waldman T, Joish V, Williamson T. Prevalence of pulmonary arterial hypertension and chronic thromboembolic pulmonary hypertension in the United States. Curr Med Res Opin. 2011 Sep;27(9):1763-8. doi: 10.1185/03007995.2011.604310. Epub 2011 Jul 27. PMID 21793646
- [Background] Delcroix M, Lang I, Pepke-Zaba J, Jansa P, D'Armini AM, Snijder R, Bresser P, Torbicki A, Mellemkjaer S, Lewczuk J, Simkova I, Barbera JA, de Perrot M, Hoeper MM, Gaine S, Speich R, Gomez-Sanchez MA, Kovacs G, Jais X, Ambroz D, Treacy C, Morsolini M, Jenkins D, Lindner J, Dartevelle P, Mayer E, Simonneau G. Long-Term Outcome of Patients With Chronic Thromboembolic Pulmonary Hypertension: Results From an International Prospective Registry. Circulation. 2016 Mar 1;133(9):859-71. doi: 10.1161/CIRCULATIONAHA.115.016522. Epub 2016 Jan 29. PMID 26826181
- [Background] Inami T, Kataoka M, Ando M, Fukuda K, Yoshino H, Satoh T. A new era of therapeutic strategies for chronic thromboembolic pulmonary hypertension by two different interventional therapies; pulmonary endarterectomy and percutaneous transluminal pulmonary angioplasty. PLoS One. 2014 Apr 11;9(4):e94587. doi: 10.1371/journal.pone.0094587. eCollection 2014. PMID 24728482
- [Background] Pepke-Zaba J, Delcroix M, Lang I, Mayer E, Jansa P, Ambroz D, Treacy C, D'Armini AM, Morsolini M, Snijder R, Bresser P, Torbicki A, Kristensen B, Lewczuk J, Simkova I, Barbera JA, de Perrot M, Hoeper MM, Gaine S, Speich R, Gomez-Sanchez MA, Kovacs G, Hamid AM, Jais X, Simonneau G. Chronic thromboembolic pulmonary hypertension (CTEPH): results from an international prospective registry. Circulation. 2011 Nov 1;124(18):1973-81. doi: 10.1161/CIRCULATIONAHA.110.015008. Epub 2011 Oct 3. PMID 21969018
- See also: a website could find all the citation above,enter the website of "https://www.ncbi.nlm.nih.gov/pubmed",input the PubMed ID of corresponding citation,and the citation will be shown in the webpage. — https://www.ncbi.nlm.nih.gov/pubmed

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT03795740/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT03795740/ICF_001.pdf